CLINICAL TRIAL: NCT01346917
Title: Prospective Randomized Controlled Study for the Effect of Intravenous Lidocaine on the Tolerability of Early Oral Feeding After Laparoscopic Colorectal Surgery in Patients With Colorectal Cancer
Brief Title: Effect of Intravenous Lidocaine on the Tolerability of Early Oral Feeding After Laparoscopic Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, HO Kim, MD, Assistant professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KHO10-1
Record Dates: First submitted 2011-04-29; First posted 2011-05-03 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Laparoscopic surgery; Postoperative ileus; Lidocaine; Early oral feeding
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Experimental)
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine — Lidocaine 1mg/kg(loading dose, just before skin incision) and lidocaine(in normal saline, total 240cc) 1mg/kg/hr with ketorolac 90mg for 24hrs.
  Arms: Lidocaine
Drug: Normal saline — Normal saline 5cc(loading dose, just before skin incision) and normal saline 240cc with ketorolac 90mg for 24hrs.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether intravenous lidocaine increase the tolerability of early oral feeding after laparoscopic colorectal surgery in patients with colorectal cancer.

* Degree of nausea/vomiting.
* Degree of postoperative pain and opioids requirement.
* Time to first flatus, time to first stool, time to tolerance of regular diet, rate of postoperative complications and duration of postoperative hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic colorectal surgery for colorectal cancer.
* Age > 18 years.
* Informed consent.

Exclusion Criteria:

* Allergy to local anesthetics.
* Severe cardiovascular, hepatic, or renal diseases.
* Pregnant or lactating patients.
* Emergency surgery.
* American Society of Anesthesiologists (ASA) class IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of postoperative nausea and vomiting. | From day of surgery to sixth postoperative day.
  Intolerance to early postoperative oral feeding is defined as the patient's having either nausea or vomiting, requiring that the patient be non-per oral status.

SECONDARY OUTCOMES:
Time to first flatus. | From day of surgery to sixth postoperative day.
Time to first passage of stool. | From day of surgery to sixth postoperative day.
Degree of postoperative pain. | From day of surgery to sixth postoperative day.
Postoperative opioid consumption. | From day of surgery to sixth postoperative day.
Time to tolerance of regular diet | From day of surgery to sixth postoperative day.
Postoperative complications | From day of surgery to thirtieth postoperative day.
Duration of postoperative hospital stay. | From day of surgery until discharge, an expected average of nine days.

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Ook Kim, M.D, Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Hyung Ook Kim, Seoul, South Korea

REFERENCES:
- [Derived] Kim HO, Lee SR, Choi WJ, Kim H. Early oral feeding following laparoscopic colorectal cancer surgery. ANZ J Surg. 2014 Jul-Aug;84(7-8):539-44. doi: 10.1111/ans.12550. Epub 2014 Feb 24. PMID 24612414